CLINICAL TRIAL: NCT00130741
Title: A Phase I, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group Study to Evaluate the Safety and Efficacy of a Combination Herbal Therapy (CHT), Versus Placebo in Improving the Overall Quality of Life and Symptoms in Patients With Irritable Bowel Syndrome (IBS)
Brief Title: Combination Herbal Therapy (CHT) Versus Placebo in Patients With Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 391-14.1.05-HMO-CTIL
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Colonic Diseases, Functional
MeSH Terms: conditions — Colonic Diseases, Functional

INTERVENTIONS:
Drug: CHT - herbal therapy

SUMMARY:
This is an 8-week double-blind, placebo-controlled, randomized, parallel-group study with an additional two week baseline observation period to evaluate the safety of combination herbal therapy (CHT) versus placebo and short and long-term efficacy in terms of improved IBS, overall quality of life (QOL) and symptomatology.

DETAILED DESCRIPTION:
Background:

IBS (Irritable Bowel Syndrome) is a disorder of motility of the entire GI tract that produces cramping, abdominal pain, constipation, and/or diarrhea and sometimes passing of mucus in bowel movements. In most people with IBS, the GI tract is highly sensitive to many stimuli, including diet and distension from gas. Among dietary suspects are high-fat or other high-calorie meals, dairy products, wheat, citrus fruits, coffee, and tea which can trigger spasms of the colon muscle. During an episode, GI tract contractions become stronger and more frequent, and the resulting rapid motility may lead to diarrhea. When colon motility is reduced, bowel movements do not occur regularly, resulting in constipation. Cramping appears to be induced by strong contractions and increased sensitivity of pain receptors in the large intestine. IBS can be triggered or intensified by stress due to communications between the central nervous system and the nervous system of the small and large intestines. This is sometimes referred to as a brain-gut connection and is supported by inspection of electroencephalogram (EEG) traces which showed significantly greater EEG abnormality in IBS patients (29.2%) than in controls (4.2%) [p<0.02]. The degree of abnormality was positively correlated with colonic motility only in IBS patients (p<0.05) allowing the authors to conclude that there is an electrophysiologic brain-gut interaction in IBS.

IBS can cause great physical discomfort and embarrassment to many of its sufferers, but is not life threatening.

There is no current consensus as to an organic cause of this syndrome and there generally appears to be no sign of disease upon physical examination except for tenderness over the large intestine. The diagnosis is symptom-based, usually through identification of the ROME II criteria for IBS. These criteria which have been accepted worldwide by clinicians and researchers as the standard for IBS diagnosis are as follows: At least 12 weeks, which need not be consecutive, in the preceding 12 months of abdominal discomfort or pain that has two of three features:

* Relieved with defecation; and/or
* Onset associated with a change in frequency of stool; and/or
* Onset associated with a change in form (appearance) of stool.

In addition the following symptoms cumulatively support the diagnosis of IBS:

* Abnormal stool frequency (for research purposes "abnormal" may be defined as >3/day and <3/week);
* Abnormal stool form (lumpy/hard or loose/ watery stool);
* Abnormal stool passage (straining, urgency, or feeling of incomplete evacuation);
* Passage of mucus;
* Bloating or feeling of abdominal distension.

The prevalence rate of IBS in 1998 in the U.S. was approximately 5,700 cases per 100,000 persons, with a much higher rate in Caucasians than in Hispanics or Afro-Americans. The total direct cost of IBS, including costs of inpatient and outpatient health services utilization and prescription medication, was greater than $1.6 billion annually in 1998 in the U.S., while the indirect costs, primarily absenteeism from work, are estimated at over $20 billion. (1 AGA: The burden of gastrointestinal diseases) IBS is treated primarily in the physician's office, with patient education, assurance and/or dietary and lifestyle modifications being the rule for mild cases, but prescription medicines being offered in more moderate cases. Prescription therapy for theses patients generally falls under two categories - drugs affecting gut physiology and psychological treatment. Very severe cases may be treated by centrally-acting agents (i.e., tricyclic antidepressants [TCAs] or selective serotonin reuptake inhibitors) together with psychological methods.

Among the medications generally used to affect gut physiology or abdominal pain are antispasmodics, tricyclic antidepressants (TCAs), loperamide, Cholestyramine (for patients with cholecystectomy or who may have idiopathic bile acid malabsorption) and serotonergic agents (5-HT3 receptor antagonists and 5-HT4 receptor agonists). These agents show relative success in improving individual symptoms only, and are only effective in specific subgroups of patients (e.g.- for diarrhea-predominant, but not constipation-predominant IBS, or visa versa). Due to the heterogeneity of IBS, an effective therapy for one may often lead to deterioration in another. For example, Alosetron, an extensively studied 5-HT3 antagonist which has shown statistically significant improvement in women with diarrhea-predominant IBS, causes constipation in 20-30% of patients, and there has been no clear evidence of a benefit for men.

There are many known side effects of anticholinergic antispasmodics and TCAs, such as: headache, dry mouth, cough, blurred vision, constipation, dysuria; postural hypotension; tachycardia, decreased libido; erectile failure; increased sensitivity to the sun; weight gain; sedation, increased sweating. Loperamide side effects include: Stomach ache, nausea, vomiting, bloating, constipation, dry mouth, drowsiness or dizziness, and cholestyramine has been known to cause constipation, heartburn, indigestion, nausea, vomiting, and stomach pain, and has caused tumors in animal studies. These profiles suggest the need for a safer, more tolerable and more comprehensive therapy for IBS.

Psychological treatments are initiated when symptoms are severe enough to impair health-related quality of life. Mental health referral may also be made for treatment of associated psychiatric disorders such as major depression. These methods include cognitive-behavioral treatment, dynamic (interpersonal) psychotherapy, hypnosis, and stress management/relaxation. Though benefit has been seen with these therapeutic methods in the relief of abdominal pain, diarrhea and anxiety, constipation has not been improved, and the effect on various subgroups of patients has not been investigated. (4 AGA Med Pos Stat)

CHT:

Some Botanical therapies, specifically combination therapies, have been tested for treatment of IBS with positive results. STW 5 (9 plant extracts) and STW 5-II (6 plant extracts) were significantly better than placebo in reducing abdominal pain and IBS symptoms after 4 weeks of therapy.

Additionally, various botanical therapies have been shown to be effective to different degrees for relief of symptoms and for improved quality of life in non-ulcer and functional dyspepsia (a condition similar to IBS). These include the following therapies tested in trials which received a rating above three in the Jadad score (a validated instrument scoring from 0-5 for assessment of clinical trial quality): celandine extract, turmeric, peppermint and caraway oils, Iberogast (peppermint leaves, caraway fruit, with or without bitter candy tuft fruit, licorice root, lemon balm leaves, angelica root, celandine herbs, milk thistle fruit and chamomile flowers), peppermint & caraway & wormwood & fennel, peppermint oil and ginger extract, artichoke leaf extract and many others with lower Jadad score ratings.

A number of herbs have been used successfully in IBS, as well. These include peppermint oil (enteric coated), globe artichoke leaf extract, and Chinese herbal medicine.

The active ingredients of CHT has been used in folklore medicine for many centuries for treatment of gastrointestinal diseases and is approved by the Israel Ministry of Health for marketing and distribution through the pharmacy . A dose toxicity test conducted in rats showed a no-observed-adverse-effect-level in male rats at doses much higher than the dose utilized in this study (measured per Kg body mass).

Considering the ethno-pharmacological and preclinical evidence for efficacy in a broad array of conditions and safety of the principal active ingredient, we, the investigators at Hadassah Medical Organization, have decided to embark upon a clinical development plan geared towards the investigation of the gastrointestinal protective and other therapeutic properties and safety of the principal active ingredient. The first study is the efficacy trial herein described.

Rationale for the study:

HCT is a new combination botanical drug substance that promises to be of value in treating various pathologies of the gastrointestinal tract, due to it's presumed "gastroprotective" and/or "gastrosynchronic" qualities. To test this hypothesis, a once daily oral dose of HCT will be self-administered to patients with IBS. The dose used is presumed to be exceptionally safe and is 37 times lower than the standard daily dose.

STUDY OBJECTIVE:

To determine the safety, tolerability and effectiveness, of 25 mg per day of HCT (20 mg principal active ingredient) compared to placebo in subjects with ROME II IBS criteria.

Basic Design Characteristics and Rationale:

This will be a double-blind, placebo-controlled, randomized, parallel group study to assess the safety and efficacy of CHT. 100 subjects with ROME II criteria IBS will provide informed consent and undergo screening procedures. Subjects fulfilling eligibility requirements will be randomized to one of the two treatment arms (will receive a subject number). After a two-week baseline observation period, and reconfirmed eligibility, subjects will be allotted enough study drug for the self administration of a daily dose of 25 mg CHT or placebo, for 4 weeks. The Week 4 clinic visit will be followed by a four week follow-up period without treatment. The day of randomization will be the week -2 visit and start of study treatment will be at the Week 0 study visit.

Throughout the study the following tools will be utilized (and variables assessed): a subject diary (for documentation of concomitant medications and concomitant medication changes and adverse events) the IBS-36 Questionnaire (for assessment of treatment-induced changes in the IBS-specific Quality of Life score), and a 6-point Likert Scale for IBS symptoms severity scoring. This tool and has been developed specifically for this study, based, in part, on similar scales in the published literature.

This early phase study is well-designed to investigate the safety and tolerability of HCT and to gain statistically significant efficacy data. The population chosen is large enough to detect a clinically significant difference in response between the active study drug and the placebo arms. The rationale for this design at such an early stage of development is based upon the recommendations of the FDA for phase I clinical studies of botanical drug substances.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-70
* Diagnosis of irritable bowel syndrome based on the following criteria (ROME II): At least 12 weeks, which need not be consecutive, in the preceding 12 months of abdominal discomfort or pain (at least once per week) with at least 2 of the following features:

  * Relief with defecation;
  * Onset associated with a change in stool frequency;
  * Onset associated with a change in stool consistency.
* At least two of the following on at least 25% of occasions or days in the last 3 months:

  * Fewer than three bowel movements a week;
  * More than three bowel movements a day;
  * Hard or lumpy stools;
  * Loose (mushy) or watery stools;
  * Straining during a bowel movement;
  * Urgency;
  * Feeling of incomplete bowel movement;
  * Passing mucus during a bowel movement;
  * Abdominal fullness, bloating or swelling.
* Women of childbearing potential must be using an acceptable method of contraception.

Exclusion Criteria:

* History of severe or intractable IBS, defined as continuous, unremitting and severe abdominal pain greater than 12 hours/day
* Concurrent diagnosis of any bowel disturbance that would interfere with the assessment or safety of the study
* History of laxative abuse
* Previous abdominal surgery (uncomplicated appendectomy, hysterectomy or cholecystectomy at least 6 months prior to entry acceptable)
* History of metabolic or inflammatory disease that may affect bowel motility, eg., inflammatory bowel disease, diabetes mellitus, sarcoidosis
* Use of the following concomitant medications: medications that can affect gastrointestinal (GI) motility; other investigational drug use (30 day "washout" required); medications affecting visceral perception; antidepressants; selective serotonin reuptake inhibitors; opioids; narcotic analgesics; antispasmodic and anticonvulsant agents; insulin or other hypoglycemic therapy; thyroid hormones; central nervous system (CNS) depressants.
* Other significant illness as determined by Investigator
* Pregnancy
* History of drug or alcohol abuse within 2 years
* Insufficient knowledge of English or Hebrew to complete self-assessments to participate in study
* Any other reason for which Investigator feels that subject's compliance is at question or safety may be compromised.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To evaluate whether CHT administered orally (PO) induces a change in the overall QOL score from baseline values at 4 weeks of treatment measured via the IBS 36 questionnaire in patients with irritable bowel syndrome, relative to placebo

SECONDARY OUTCOMES:
30% change on the IBS-36 from baseline to 4 weeks ("no" or "yes")
Change on IBS-36 from 4 weeks (last treatment taken) and 8 weeks (i.e., after 4 weeks of "washout")
Change in IBS symptoms severity score from baseline to 4 weeks
Change in IBS symptoms severity score from 4 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel